CLINICAL TRIAL: NCT03725930
Title: Premedication by Clonidine Intranasal in Pediatric Surgery
Acronym: CLONIPREM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016_37; 2017-003638-10 (EudraCT Number)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Child Preschool
Keywords: paediatric; premedication; clonidine; intranasal
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clonidine (Active Comparator): This arm will receive intra nasal Clonidine as a premedication before surgery
  Interventions: Drug: Clonidine
- Placebo (Placebo Comparator): This arm will receive intra nasal Placebo as a premedication before surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clonidine — clonidine intranasal premedication in preschool infants
  Arms: Clonidine
Other: Placebo — Placebo intranasal premedication
  Arms: Placebo

SUMMARY:
There are few studies using intra nasal way to dispense premedication in pediatrics.

This study will evaluate anxiolysis effect of Intranasal premedication with Clonidine vs Placebo.

Two groups, randomized,

Total of 150 patients (75 in each group) :

Involvement in study for one patient : 7 days Duration of study including inclusion and data analysis : 18 months (inclusion 12 months; data analysis 6 months)

ELIGIBILITY:
Inclusion Criteria:

1. Child from 1 to 5 years
2. Weight between 10 to 25 kgs
3. Scheduled minor surgery
4. Oral and written information and consent given by main investigator to both of the parents or legal(s) representative(s).
5. ASA score 1 or 2
6. Patient with social care insurance

Exclusion Criteria:

1. Refusal of one of the parental authority or legal representing
2. Concomitant participation to a clinical trial with use of a drug
3. Known hypersensitivity or contraindication to Clonidine or one of its excipients
4. Airway infection within 3 weeks before inclusion
5. Intravenous induction of anesthesia
6. Antecedent of arrhythmia or congenital heart disease
7. Mental disorder or current psychoactive medication

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Anxiolysis score | at 30 minutes after premedication
  Anxiolysis score (1 : Anxious, crying; 2 : Anxious; 3 : Calm, not cooperative; 4 : Calm, cooperative

SECONDARY OUTCOMES:
Acceptation of mask at the induction of anesthesia | 1 hour after premedication
  Yes / No
Agitation score after the extubation | 15 min after extubation
  Agitation score : 0 : Patient

CONTACTS AND LOCATIONS:
Overall Officials: Dina BERT, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU Lille, Lille, Nord, France